CLINICAL TRIAL: NCT03099369
Title: The Effectiveness of Daily Step-based Exercise Therapy Using Fitness Monitors for Peripheral Artery Disease: The EASY FIT Trial
Brief Title: Daily Step-based Exercise Using Fitness Monitors for Peripheral Artery Disease
Acronym: EASY FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-3427
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-03

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Peripheral Arterial Disease; Exercise; Step Count; Fitness Monitor; Mobile Health; Walking Ability; Quality of Life
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Step-based Exercise Group (Experimental): The experimental group will receive the following 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day (based on evidence that at least 5,000 a day is associated with better health). The Fitbit Fitness Monitor used for tracking.
  * Week 1: walk at least 3,000 steps every day.
  * Week 2: walk at least 3,500 steps every day.
  * Week 3: walk at least 4,000 steps every day.
  * Week 4: walk at least 4,500 steps every day.
  * Weeks 5-12: walk at least 5,000 steps every day.
  Interventions: Behavioral: Daily Step-based Exercise; Other: Fitbit Fitness Monitor
- Symptom-based Exercise Group (Active Comparator): The active comparator group (ie. control group) will receive the following 12-week symptom-based exercise prescription (adapted from practice guidelines).
  * Walk on a flat surface at a constant speed until there is mild to moderate pain
  * Rest until the pain has completely ceased
  * Resume walking at the same speed
  * Increase the speed when you can walk 8 minutes without stopping for leg symptoms
  * Continue this exercise routine for 45 consecutive minutes, 3 to 5 days a week.
  Interventions: Behavioral: Symptom-based Exercise; Other: Fitbit Fitness Monitor

INTERVENTIONS:
Behavioral: Daily Step-based Exercise — A 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day.
  Arms: Daily Step-based Exercise Group
Behavioral: Symptom-based Exercise — A 12-week symptom-based exercise prescription adapted from clinical practice guidelines.
  Arms: Symptom-based Exercise Group
Other: Fitbit Fitness Monitor — Used by the experimental group to assess outcome and to guide exercise therapy; used by the active comparator group to assess outcome only

SUMMARY:
Peripheral artery disease (PAD) is caused by blockages in the leg arteries. PAD limits patients' walking ability and quality of life. For patients with PAD, home exercise programs can improve walking ability and quality of life. In many patient populations, walking more than 5,000 steps a day is associated with better health. Currently, the benefit of walking more than 5,000 steps a day in patients with PAD has not been well studied.

The purpose of this clinical trial is to compare two different home exercise programs in patients with PAD: walking at least 5,000 steps a day with the help of fitness monitors vs. walking 45 consecutive minutes for 3 to 5 days a week (a common exercise prescription for PAD). This study has the potential to demonstrate that, with the help of fitness monitors, walking at least 5,000 steps a day can improve walking ability and quality of life for patients with PAD.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is the third leading cause of cardiovascular morbidity, following coronary artery disease and stroke. Symptoms of PAD include claudication, decreased exercise capacity, progressive functional impairment, and decreased quality of life. Structured exercise therapy is a cornerstone of treating symptomatic PAD. Guidelines recommend a symptom-based exercise program that uses claudication to moderate walking sessions.

Home exercise programs have demonstrated efficacy in improving walking ability and quality of life for symptomatic PAD patients. In the general population and patients with certain chronic diseases, walking more than 5,000 steps a day has been associated with better health. The efficacy of walking more than 5,000 steps a day has not been well studied in symptomatic PAD patients.

The EASY FIT Trial is a single-center prospective randomized controlled trial comparing the effectiveness of a daily step-based exercise program (walking at least 5,000 steps a day) vs. a guideline-recommended symptom-based exercise program (walking 45 consecutive minutes for 3 to 5 days a week), on improving walking ability and quality of life in patients with symptomatic PAD. The study will enroll and randomize 40 patients with symptomatic PAD (20 to each exercise program).The results of this study have the potential to create an effective, safe, feasible, and sustainable exercise program that can help PAD patients have greater walking ability and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Diagnosis of lower extremity PAD based on at least 1 of the following criteria:

  * Ankle-brachial index (ABI) of 0.9 or less in one or both legs
  * Invasive angiography demonstrating obstructive lower extremity artery disease
  * Endovascular or surgical revascularization of lower extremity artery
* Symptomatic lower extremity PAD, characterized by 1 of the following:

  * Fontaine Stage IIa: intermittent claudication after walking > 200 meters
  * Fontaine Stage IIb: intermittent claudication after walking < 200 meters
* Have the availability of a suitable environment in which to walk
* Have a mobile phone with WiFi and Bluetooth capability
* Have the ability to read and speak the English language

Exclusion Criteria:

* Wheelchair bound
* Use of a walking aid (ie. cane, crutches, walker, motorized chair)
* Below or above the knee amputation
* Leg pain at rest
* Acute or critical limb ischemia
* Ischemic ulceration or gangrene
* Diabetes mellitus complicated by neuropathy
* Walking impairment due to another cause than PAD
* Ongoing evaluation for coronary artery disease (ie. awaiting a stress test or cardiac catheterization)
* Active coronary artery disease requiring the initiation or uptitration of an anti-anginal medication
* Angina with Canadian Cardiovascular Society (CCS) class 3-4 symptoms
* Myocardial infarction in the last 3 months
* Active congestive heart failure requiring the initiation or uptitration of diuretic therapy
* Congestive heart failure with New York Heart Association (NYHA) class 3-4 symptoms
* Active arrhythmia requiring the initiation or uptitration of an anti-arrhythmic medication
* Severe valve disease
* Active cancer or malignancy (not in remission)
* End-stage renal disease requiring hemodialysis or peritoneal dialysis
* Advanced liver disease, defined as cirrhosis
* Thyroid disease with abnormal TSH in the past 3 months
* Severe cognitive dysfunction, defined as dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Lee, MD, Principal Investigator — University of North Carolina; Prashant Kaul, MD, Principal Investigator — University of North Carolina; George A Stouffer, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily Step-based Exercise Group: The experimental group will receive the following 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day (based on evidence that at least 5,000 a day is associated with better health). The Fitbit Fitness Monitor will be used for tracking.
  * Week 1: walk at least 3,000 steps every day.
  * Week 2: walk at least 3,500 steps every day.
  * Week 3: walk at least 4,000 steps every day.
  * Week 4: walk at least 4,500 steps every day.
  * Weeks 5-12: walk at least 5,000 steps every day.
  Daily Step-based Exercise: A 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day.
  Fitbit Fitness Monitor: Used by the experimental group to assess outcome and to guide exercise therapy; used by the active comparator group to assess outcome only
- Symptom-based Exercise Group: The active comparator group (i.e., control group) will receive the following 12-week symptom-based exercise prescription (adapted from practice guidelines).
  * Walk on a flat surface at a constant speed until there is mild to moderate pain
  * Rest until the pain has completely ceased
  * Resume walking at the same speed
  * Increase the speed when you can walk 8 minutes without stopping for leg symptoms
  * Continue this exercise routine for 45 consecutive minutes, 3 to 5 days a week.
  Symptom-based Exercise: A 12-week symptom-based exercise prescription adapted from clinical practice guidelines.
  Fitbit Fitness Monitor: Used by the experimental group to assess outcome and to guide exercise therapy; used by the active comparator group to assess outcome only
Period: Overall Study
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group
Started | 11 | 9
Completed | 5 | 5
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.5) | 58.6 (16.5) | 60.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Daily Walking Distance Over 7 Consecutive Days
Description: At baseline, both groups will be instructed to wear their fitness monitors for 7 consecutive days. After 3 months of the exercise program, both groups will be instructed to wear their fitness monitors for 7 consecutive days. During each 7-day period, all patients will be instructed to walk continuously for at least one extended period of time on a daily basis. Given that this is a pilot study, the duration and frequency of these extended periods of time will be at the patients' discretion. The change in the mean daily walking distance at 3 months will be the primary outcome.
Time Frame: Baseline, Month 3
Population: Data were not collected for 10 participants because of their inability to complete prescribed exercise program or to upload Fitbit data.
Measure: Mean (Standard Deviation); unit: steps
Groups:
- Daily Step-based Exercise Group: The experimental group will receive the following 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day (based on evidence that at least 5,000 a day is associated with better health). The Fitbit Fitness Monitor used for tracking.
  * Week 1: walk at least 3,000 steps every day.
  * Week 2: walk at least 3,500 steps every day.
  * Week 3: walk at least 4,000 steps every day.
  * Week 4: walk at least 4,500 steps every day.
  * Weeks 5-12: walk at least 5,000 steps every day.
  Daily Step-based Exercise: A 12-week step-based exercise prescription with the eventual goal of walking at least 5,000 steps a day.
  Fitbit Fitness Monitor: Used by the experimental group to assess outcome and to guide exercise therapy; used by the active comparator group to assess outcome only
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group
Number analyzed (Participants) | 5 | 5
steps | 754.2 (1621.7) | -1160 (2963.2)

2. Secondary Outcome: Change in the Peripheral Artery Questionnaire (PAQ) Summary Score
Description: At baseline, both groups will be asked to complete the Peripheral Artery Questionnaire (PAQ), which is a quality-of-life survey with a summary score ranging from 0 to 100 (with 100 indicating the highest quality of life). After 3 months of the exercise program, both groups will be asked to complete the PAQ again. The change in the summary score at 3 months will the secondary outcome.
Time Frame: Baseline, Month 3
Population: None of the participants could be reached to obtain both baseline and endpoint telephone survey data. Therefore, data for this outcome measure are unavailable.
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in the Vascular Quality of Life Questionnaire (VascuQol) Summary Score
Description: At baseline, both groups will be asked to complete the Vascular Quality of Life Questionnaire (VascuQol), which is a quality-of-life survey with a summary score ranging from 25 to 175 (with 175 indicating the highest quality of life). After 3 months of the exercise program, both groups will be asked to complete the VascuQol survey again. The change in the summary score at 3 months will the secondary outcome.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected based on participant chart review during the baseline assessment period (1 week), the 12-week intervention period, and the final assessment period (1 week), for a total of approximately 14 weeks.
Arm/Group | Daily Step-based Exercise Group | Symptom-based Exercise Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03099369/Prot_SAP_000.pdf